CLINICAL TRIAL: NCT07344207
Title: A Prospective, Open-Label, Randomized Controlled Trial of an Artificial Intelligence Enabled Electrocardiography System for Preoperative Detection of Pulmonary Hypertension and Related Diseases(GUARD-PH)
Brief Title: GUARD-PH: Guided Use of AI-ECG for Risk Detection of PH in Surgery (GUARD-PH Trial)
Acronym: GUARD-PH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-10-004CCF
Record Dates: First submitted 2025-12-21; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hypertension (Diagnosis); Pre-operative Assessment; Postoperative Complications (Cardiopulmonary); Treatment Outcomes
Keywords: Artificial Intelligence; Electrocardiography; AI-ECG; Preoperative Detection; Screening
MeSH Terms: conditions — Hypertension, Pulmonary; Disease; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-ECG Screening Group (Experimental): The physician responsible for the participant in this arm will receive the results generated by the artificial intelligence-enabled electrocardiography (AI-ECG) system for pulmonary hypertension.
  Interventions: Diagnostic Test: Artificial Intelligence-Enabled Electrocardiography System
- Standard of Care Group (No Intervention): The physician responsible for the participant in this arm will not receive the results generated by the artificial intelligence-enabled electrocardiography (AI-ECG) system for pulmonary hypertension.

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence-Enabled Electrocardiography System — The intervention involves using an artificial intelligence-enabled electrocardiography system to analyze standard ECGs for the preoperative detection of pulmonary hypertension.
  Arms: AI-ECG Screening Group

SUMMARY:
This study is a prospective, open-label, randomized controlled trial designed to evaluate a new artificial intelligence (AI) tool for heart monitoring. Researchers will use an AI-enabled electrocardiography (ECG) system to screen patients before they undergo surgery. The main goal is to determine if this AI system can accurately detect pulmonary hypertension and related heart diseases in the preoperative setting. The study is being conducted at Taipei Veterans General Hospital.

DETAILED DESCRIPTION:
This is an open-label, prospective, randomized controlled trial at Taipei Veterans General Hospital. Approximately 1,380 adult patients who already have a preoperative electrocardiogram (ECG) scheduled as part of routine care and have an established plan for elective surgery will be enrolled, along with approximately 30-60 participating physicians responsible for preoperative assessment and perioperative clinical care. The study evaluates whether integrating the Taiwan Medical Imaging Pulmonary Hypertension Detection System (TAIMedImg PHDS), an ECG-based clinical decision-support tool, during the preoperative preparation period can enable earlier identification of patients at risk of pulmonary hypertension and cardiopulmonary complications, and supports assessment of the potential cost-effectiveness of earlier risk recognition.

Patients are randomized to determine whether their responsible participating physician will receive TAIMedImg PHDS output derived from the patient's routine ECG. In the intervention arm, research staff upload the ECG to TAIMedImg PHDS and provide the analysis result to the participating physician; all other processes proceed as usual care. In the control arm, usual care proceeds without provision of TAIMedImg PHDS output. Randomization affects only access to this supplementary ECG-based output; it does not change patients' scheduled tests, clinical workflow, or rights to care. Clinical evaluation and management remain at the physician's discretion according to standard practice.

The study measures physicians' responses to ECG interpretation with versus without TAIMedImg PHDS output and documents the clinical decision-making trajectory, using routinely available medical record data for analysis. Results may inform improved preoperative pulmonary hypertension risk assessment and future perioperative care.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years.
2. Patients scheduled for non-cardiac surgery under general anesthesia.
3. Patients who have a scheduled standard preoperative electrocardiogram (ECG).
4. Patients capable of understanding the study and willing to provide medical records for research purposes, and who have signed the informed consent form.

Exclusion Criteria:

1. Patients scheduled for emergency surgery.
2. Patients who explicitly refuse to participate or withdraw consent.
3. Patients with specific comorbidities that interfere with ECG interpretation or data collection (e.g., implanted pacemakers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
The incidence of newly diagnosed pulmonary hypertension or pulmonary hypertension-related cardiopulmonary diseases | Before surgery, or within 90 days after electrocardiography in patients who did not undergo surgery.
  The incidence of newly diagnosed pulmonary hypertension (defined as an echocardiographic right ventricular systolic pressure > 50 mmHg) or pulmonary hypertension-related cardiopulmonary diseases before surgery, or within 90 days after electrocardiography in patients who did not undergo surgery.

SECONDARY OUTCOMES:
Incidence of Surgical Complications | From the date of surgery up to 3 months post-operation.
  Comparison of the incidence rates of surgical complications between the two groups.
Length of Hospital Stay | From admission until hospital discharge (assessed up to 3 months).
  Comparison of the total duration of hospitalization (in days) between the intervention and control groups.
Cardiovascular Mortality | From the date of surgery up to 3 months post-operation.
  Evaluation of the rates of cardiovascular-related death between the two groups during the postoperative observation period.
All-Cause Mortality | From the date of surgery up to 3 months post-operation.
  Evaluation of the rates of all cause mortality between the two groups during the postoperative observation period.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT07344207/Prot_SAP_000.pdf